CLINICAL TRIAL: NCT07044154
Title: Effect of Sun Tai Chi on the Cardiopulmonary System and Mental Health in University Students: A Mixed Randomized Clinical Trial
Brief Title: Effect of Sun Tai Chi on the Cardiopulmonary System and Mental Health in University Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Pamela Ling Campos Rojas, kinesiologist, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90/2025
Record Dates: First submitted 2025-06-12; First posted 2025-06-29 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Mental Health Conditions; University Students
Keywords: university students; Sun Tai Chi; cardiac autonomic modulation; cardiopulmonary capacity; mental health; qualitative perception
MeSH Terms: conditions — Psychological Well-Being | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be conducted, using a mixed quantitative-qualitative phenomenological design, single-blind, prospective longitudinal, with non-probabilistic convenience sampling. First, the quantitative phase will be carried out, followed by the qualitative phase.
  Once the Tai Chi intervention is completed (beginning one week after the final session), the qualitative phase will begin.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Sun Tai Chi Group (Experimental): The group will participate in 60-minute Sun Tai Chi sessions, held twice per week over a 12-week period.
  Interventions: Other: Tai Chi (Sun Style)
- Control (Other): The group will receive informational material on healthy lifestyle topics and will not receive the Sun Tai Chi intervention.
  Interventions: Behavioral: Health lifestyle education

INTERVENTIONS:
Other: Tai Chi (Sun Style) — The Sun Tai Chi intervention will be conducted by a Sun Tai Chi instructor with 7 years of teaching experience and will take place in an exercise room at the Catholic University of Maule. The intervention will last for 12 weeks, with a frequency of twice per week, and each class will last 60 minutes. Each session will begin with 10 minutes of warm-up exercises, followed by 20 minutes of basic Sun Tai Chi exercises, including lower limb movements, overall body mobility at a slow pace, precise movements of the hands and feet, and proper body alignment. This will be followed by 20 minutes of practice of the basic movement sequence of Sun Tai Chi (Taolú), and will conclude with 5 minutes of meditation and 5 minutes of relaxation exercises.
  Arms: Experimental: Sun Tai Chi Group
Behavioral: Health lifestyle education — The control group will receive guidance on a healthy physical and mental lifestyle.
  Arms: Control

SUMMARY:
Currently, university students face physical and mental health issues, which are reflected in low levels of physical activity, a decline in healthy eating behaviors, and a high prevalence of mental health symptoms such as stress, anxiety, and depression. Therefore, it is necessary to develop safe, effective, and sustainable interventions that support comprehensive health and provide formative experiences that reinforce the importance of developing healthy lifestyle habits and self-care.

In this regard, Tai Chi has been shown to offer physical and mental health benefits. Tai Chi is a low- to moderate-intensity exercise with low joint impact, which facilitates the transition from a sedentary to an active lifestyle.

Considering the health problems experienced by university students, it is proposed that a Tai Chi intervention could help produce beneficial effects on both physical and mental health. In this context, the present study aims to implement Tai Chi classes with the objective of determining their effect on the cardiac autonomic system, mental health, and the perception of benefits, facilitators, and barriers among participating university students compared to a control group.

DETAILED DESCRIPTION:
In Chile, there are currently over 1.2 million undergraduate university students who exhibit low levels of physical activity and mental health issues such as anxiety and depression. These problems tend to worsen after the first year of higher education, along with the development of unhealthy eating habits and weight gain.

In this context, Tai Chi has shown multiple benefits for overall health. Specifically, the Sun style of Tai Chi is characterized by gentle and accessible movements, making it well-suited to the university setting, and has demonstrated positive effects on both physical and mental health.

Previous studies indicate that regular practice of Tai Chi may positively influence autonomic cardiac control, measured through heart rate variability (HRV), as well as mental health. However, the available evidence is still limited and heterogeneous.

This study aims to evaluate, in university students, the effects of a 12-week Sun Tai Chi program, with 60-minute sessions held twice per week, on the following:

* Heart Rate Variability (HRV), as a marker of cardiovascular health and stress,
* Mental health, assessed with the Depression Anxiety Stress Scales - 21 Items (DASS-21 scale),
* Participants' qualitative perceptions regarding the program's benefits, barriers, and facilitators.

Given the limited research on Tai Chi in university student populations, this study seeks to contribute evidence on its potential comprehensive health benefits in this group.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate university students
* Aged 18 to 29 years
* Both sexes
* Present mental health symptoms assessed by the Depression Anxiety Stress Scales - 21 Items (DASS-21) questionnaire, according to cutoff points established by Lovibond et al., ranging from mild to severe in any of the subscales of stress (score 15 to 33), anxiety (score 8 to 19), or depression (score 10 to 27).
* Report a healthy physical condition suitable for Tai Chi practice (self-reported).

Exclusion Criteria:

* Engage in a high level of physical activity according to the International Physical Activity Questionnaire (IPAQ) or have regularly practiced moderate to high intensity physical activity in the last 3 months.
* Report chronic illnesses that limit or contraindicate the practice of exercises required in Tai Chi.
* Present cardiovascular, pulmonary, or neurological diseases.
* Exhibit either no mental health impairment or severe impairment according to cutoff scores established by Lovibond et al. in the DASS-21 questionnaire (stress subscale score equal to or greater than 14 or equal to or less than 37, anxiety subscale score equal to or greater than 7 or equal to or less than 20, depression subscale score equal to or greater than 9 or equal to or less than 28).
* Present specific psychiatric diagnoses, such as Attention-Deficit/Hyperactivity Disorder (ADHD), self-reported during the initial telephone interview.
* Consume medications for mental health treatment.
* Consume medications or substances that influence cardiac autonomic modulation (e.g., beta-blockers).

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
DASS-21 stress | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  Stress will be measured using the stress subdomain of the DASS-21, which ranges from 0 to 21 points, with higher scores indicating higher levels of stress.
DASS-21 anxiety | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  Anxiety will be measured using the anxiety subdomain of the DASS-21, which ranges from 0 to 21 points, with higher scores indicating higher levels of anxiety.
DASS-21 depression | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  Depression will be measured using the depression subdomain of the DASS-21, which ranges from 0 to 21 points, with higher scores indicating higher levels of depression.
RMSSD | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  RMSSD (ms) is an index of parasympathetic cardiac autonomic modulation derived from the analysis of RR intervals (iRR).
SDNN | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  SDNN (ms) is an index of overall heart rate variability reflecting the cardiac autonomic modulation derived from the analysis of RR intervals (iRR).
Low frequency (LF) | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  LF (ms2) is an index of parasympathetic and sympathetic cardiac autonomic modulation derived from the analysis of RR intervals (iRR).
High frequency (HF) | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  HF (ms2) is an index of parasympathetic cardiac autonomic modulation derived from the analysis of RR intervals (iRR).
Low frequency/Hight frequency ratio (LF/HF) | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  LF/HF is an index reflecting the balance between the parasympathetic and sympathetic cardiac autonomic modulation derived from the analysis of RR intervals (iRR).
Pattern with no variation (0V) | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  0V (%) is a pattern quantified through symbolic analyses of the RR intervals (iRR) reflecting the sympathetic cardiac modulation.
Pattern with two unlike variation (2ULV) | Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  2ULV (%) is a pattern quantified through symbolic analyses of the RR intervals (iRR) reflecting the parasympathetic cardiac modulation.
Baroreflex sensitivity (BRS) | Time Frame: Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  Baroreflex sensitivity is an index that assesses the heart rate response to changes in blood pressure and serves as an indicator of cardiovascular health.
LFSAP | Time Frame: Initial evaluation: Prior to the intervention (week 0) Intermediate evaluation: After 6 weeks of intervention Final evaluation: After 12 weeks of intervention
  The low-frequency index of systolic arterial pressure (LFSAP) reflects the vascular sympathetic autonomic modulation.
Qualitative perception | It will be conducted one week after the last Tai Chi class.
  The qualitative perception of the participants will consider the perceived benefits, barriers, and facilitators. Data will be collected through semi-structured interviews and focus groups, using a qualitative approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica del Maule, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No